CLINICAL TRIAL: NCT05810506
Title: Evaluation of Anthropometric Measurements and Biochemical Parameters in Non-Alcoholic Fatty Liver Patients and Healthy Individuals
Brief Title: Non-Alcoholic Fatty Liver Disease and Anthropometric Measurements
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Tuba ONAY, Research Assistant Doctor /Principal İnvestigator, Bandırma Onyedi Eylül University
Other Study IDs: Tuba ONAY
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver disease; anthropometric measurements; body shape index; body roundness index; visceral adiposity index
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Healthy individuals; they were required to sign the voluntary consent form, not consume alcohol, be between 30-64 years old, and not have any acute or chronic diseases. Individuals outside these criteria were not included in the study. In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention.
  Interventions: Other: In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention.
- NAFLD: NAFLD patients included in the study should sign a voluntary consent form, do not consume alcohol, be between 30-64 years old, have been diagnosed with NAFLD by applying to the gastroenterology outpatient clinic, have no other diseases, and should not use medication. In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention.
  Interventions: Other: In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention.

INTERVENTIONS:
Other: In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention. — In the study, biochemical parameters will be taken from the anthropometric measurements and files of the patients without any intervention.

SUMMARY:
The aim of this study; Which anthropometric measurement and ratio (BMI, waist circumference, hip circumference, waist-to-hip ratio, neck circumference, waist-height ratio, body shape index, body roundness index, visceral adiposity index) is a better indicator in healthy individuals with NAFLD and their biochemical parameters is to evaluate.

DETAILED DESCRIPTION:
NAFLD patients included in the study should sign a voluntary consent form, do not consume alcohol, be between 30-64 years old, have been diagnosed with NAFLD by applying to the gastroenterology outpatient clinic, have no other diseases, and should not use medication. Healthy individuals; they were required to sign the voluntary consent form, not consume alcohol, be between 30-64 years old, and not have any acute or chronic diseases. Individuals outside these criteria were not included in the study. The reason for the 30-64 age limit for individuals with NAFLD in the study is that NAFLD is more common in this age group. The same criteria were also taken into account in healthy individuals to avoid differences between groups. Individuals who met the inclusion criteria of the study and accepted to participate in the study voluntarily were selected by random sampling method and the sample of the study was formed. For the study, research permission was obtained from Gülhane Training and Research Hospital and ethical approval of the study from Ankara University Ethics Committee (56786525-050.04.04/236883). Written and verbal consent was obtained from the patients before starting the study. The research was conducted in accordance with both the Declarations of Helsinki and Istanbul. Biochemical Parameters Fasting blood glucose, total cholesterol, triglyceride, HDL, VLDL, LDL, ALP, AST, ALT and GGT values of the individuals participating in the study were obtained from the files with the permission of the patients.

Anthropometric Measurements The data were collected using a questionnaire form and face-to-face interview method. In the study, individuals' body weight (kg), height (cm), waist circumference (cm), hip circumference (cm), neck circumference (cm) measurements were taken in accordance with the method, and these measurement values were used to measure BMI, waist-height ratio, waist-hip ratio, body composition (fat mass, muscle mass, etc.), body shape index, body roundness index, visceral adiposity index measurements were calculated. Body mass index was calculated by dividing the body weight by the square of the height. Other anthropometric measurements and ratios were calculated using appropriate formulas.

ELIGIBILITY:
Inclusion Criteria for NAFLD patients:

* should sign a voluntary consent form
* do not consume alcohol
* be between 30-64 years old
* have been diagnosed with NAFLD by applying to the gastroenterology outpatient clinic
* have no other diseases
* should not use medication

Inclusion Criteria for healthy individuals:

* should sign a voluntary consent form
* do not consume alcohol
* be between 30-64 years old
* not have any acute or chronic diseases

Exclusion Criteria for NAFLD patients:

* consuming alcohol
* not be between 30-64 years old
* being pregnant or lactating
* any surgery in the last 3 months
* Not being diagnosed with NAFLD
* Hepatitis B-C, Wilson's disease, autoimmune liver diseases, cancer, cirrhosis, inflammatory bowel diseases, celiac, diabetes, cystic fibrosis, hereditary diseases, irritable bowel syndrome, kidney diseases, AIDS-HIV etc. have a disease
* using any medication other than fatty liver

Exclusion Criteria for healthy individuals:

* consuming alcohol
* any acute or chronic illness
* being pregnant-lactating
* using any medicine
* not be between 30-64 years old

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals with non-alcoholic fatty liver disease
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Body weight | Six month
  Body weight measurements of the patients will be made by removing thick clothes and shoes, and by means of TANITA BC-418 MA brand Bioelectrical Impedance Analysis (BIA).
Height | Six month
  The height of the patients will be measured with a stadiometer while the feet are together and the head is in the Frankford plane.
Body fat percentage | Six month
  The body fat mass of individuals will be measured with the TANITA BC-418 MA BIA analyzer.
Neck circumference | Six month
  Measure with a non-stretchable tape measure horizontally at the upper edge of the laryngeal prominence with the head upright and eyes facing forward.
Waist circumference | Six month
  The patient's side will be passed to the side of the patient and the circumference passing through the middle point will be measured between the lowest point of the rib bone and the iliac crest.
Hip circumference | Six month
  The largest circumference between the waist and knees will be measured by going to the side of the patient.
Body mass index | Six month
  It will be calculated by dividing the body weight by the square of the height
Waist-to-length ratio | Six month
  It is the ratio of waist circumference to height.
Waist to hip ratio | Six month
  It is the ratio of waist circumference to hip circumference.
Body shape index | Six month
  Body shape index of patients; with height, waist circumference and BMI values; It will be calculated using the formula [Waist circumference/ (BKİ )2/3* Height 1/2].
Body roundness index | Six month
  The body roundness index of the patients will be calculated using the formula [364.2-365.5x√1-[(waist circumference/(2π))2/(0.5 x height)2].
Visceral adiposity index | Six month
  Patients' visceral adiposity index for men: [Waist circumference/ 39.68 + (1.88 × [BMI])] × [(TG)/1.03] × (1.31/HDL); for women: will be calculated using the formulas [Waist circumference /36.58 + (1.89 × BMI)] × (TG/0.81) × (1.52/HDL).

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma onyedi eylül unıversıty, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not planned.